CLINICAL TRIAL: NCT03282604
Title: The Ideal Length of the Nasotracheal Tube Considering Nasotracheal Tube Size
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2017-0048
Record Dates: First submitted 2017-09-11; First posted 2017-09-14 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Nasotracheal Intubation for General Anesthesia
Keywords: Intubation; Intratracheal; Nasopharynx

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- male
- female

SUMMARY:
The nasotracheal intubation is preferred for oral surgery; it provides an easier view of the surgical field. However, nasotracheal tubes are produced by foreign countries. Tubes are often not fitted in anatomy of Korean people because of small nostril. When the size of the tube is chosen by nostril size, the length of nasotracheal tube is not appropriate to the glottis. The aim of this study is to evaluate the appropriateness of the tube depth and to suggest the ideal length of the nasotracheal tube during the intubation of the selected tracheal tube in consideration of the size of the nasal cavity in Koreans. 146 patients (73 males and 73 females) who are scheduled for nasal intubation for general anesthesia will be enrolled. The primary outcome is the ideal length of tube that allows the distance from the vocal cords to the proximal portion of the tube cuff to be greater than 2 cm and the tip of the intubated tube to be located 5 ± 2 cm above the tracheal carina. The size of nostril, length from the nare to the carina and vocal cord are measured.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are scheduled for nasotracheal intubation for general anesthesia

Exclusion Criteria:

1. age<20 years
2. ASA class III or more
3. pregnancy
4. emergency surgery
5. nasal airway disease
6. expected difficult intubation (difficult intubation history, Modified Mallampati score 4, mouth opening <2cm, facial anomaly)
7. cervical movement disorder (cervical disease, cervical pain)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for nasotracheal intubation for general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
the ideal length of the nasotracheal tube during the intubation of the selected tracheal tube in consideration of the size of the nasal cavity in Koreans | through study completion, an average of 1 year
  the ideal length of tube that allows the distance from the vocal cords to the proximal portion of the tube cuff to be greater than 2 cm and the tip of the intubated tube to be located 5 ± 2 cm above the tracheal carina.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stoneham MD. The nasopharyngeal airway. Assessment of position by fibreoptic laryngoscopy. Anaesthesia. 1993 Jul;48(7):575-80. doi: 10.1111/j.1365-2044.1993.tb07119.x. PMID 8346770
- [Background] Reed DB, Clinton JE. Proper depth of placement of nasotracheal tubes in adults prior to radiographic confirmation. Acad Emerg Med. 1997 Dec;4(12):1111-4. doi: 10.1111/j.1553-2712.1997.tb03691.x. PMID 9408424
- [Background] Han DW, Shim YH, Shin CS, Lee YW, Lee JS, Ahn SW. Estimation of the length of the nares-vocal cord. Anesth Analg. 2005 May;100(5):1533-1535. doi: 10.1213/01.ANE.0000149900.68354.33. PMID 15845720